CLINICAL TRIAL: NCT04462120
Title: Association Between IL-12RB and TNF-alpha Gene Polymorphism With Susceptibility and Progress of Covid-19 SARS-CoV-2: A Case Control Study
Brief Title: IL-12RB and TNF-alpha Gene Polymorphism and Susceptibility and Progress of Covid-19 SARS-CoV-2: A Case Control Study
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Aliae AR Mohamed Hussein, Professor of Pulmonology, Assiut University
Other Study IDs: AssiutU15
Record Dates: First submitted 2020-06-19; First posted 2020-07-08 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2020-07

CONDITIONS: Covid-19
Keywords: COVID-19; corona virus disease; SARS-CoV-2; IL-12 RB gene polymorphism; TNF gene polymorphism
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A novel coronavirus was identified in late 2019 in Wuhan, China On 11 February, The International Committee on Taxonomy of Viruses (ICTV) announced that the official classification of the new coronavirus (2019-nCoV) is called severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2). The World Health Organization (WHO) announced on the same day that the official name of the disease caused by the virus is Corona Virus Disease-19 (COVID-19). WHO has declared the infection a Pandemic on March 11, 2020. Based on previous studies on SARS in 2003 and SARS-MERS 2013 there was a genetic polymorphism associated with the susceptibility and severity of the disease.

Interleukin-12 (IL-12) is a cytokine secreted by activated phagocytes and dendritic cells. It plays a pivotal role in promoting Th1-type immune responses and cell-mediated immunity. IL-12 triggers many biological functions: it stimulates the proliferation of activated T- and NK-cells, enhances T- and NK-cell-mediated cytolytic activity, and induces the production of IFN-γ by both T-and NK-cells. The interferon-γ production induced by IL-12 forms a major link between innate and adaptive immunity. A recent study revealed that interferon-mediated immunopathological events are associated with atypical innate and adaptive immune responses in SARS patients.

Also, TNF-α is a key mediator of the inflammatory response and is critical for host defense against a wide variety of pathogenic microbes. However, the over-expression of this cytokine may lead to badness in disease recovery. The dual role of TNF, acting as an agent of both innate immunity and inflammatory pathology, poses a considerable challenge for gene regulation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with confirmed COVID-19 PCR ( mild, moderate and severe cases) admitted to wards or ICU Assiut University Hospitals

Exclusion Criteria:

* Suspected or non confirmed cases of COVID-19

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with confirmed COVID-19 PCR ( mild, moderate and severe cases) admitted to wards or ICU Assiut University Hospitals
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-06-16 (Actual); Primary Completion 2020-06-18 (Actual); Study Completion 2020-07-30 (Estimated)

PRIMARY OUTCOMES:
Measure level of polymorphisms of interleukin (IL)-12 receptor B1 (IL-12RB1) and TNF- α alpha on COVID-19 related severe acute respiratory syndrome (SARS-CoV-2). | day 1
  genetic polymorphism

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - AssiutU, Asyut
  - Assiut University Hospitals, Asyut

IPD SHARING:
Plan to Share IPD: No